CLINICAL TRIAL: NCT00916058
Title: A Phase 1-2 Study of a Novel Conditioning Regimen of Bendamustine and Melphalan Followed by Autologous Stem Cell Transplant for Patients With Multiple Myeloma
Brief Title: Conditioning Regimen of Bendamustine and Melphalan Followed by Transplant in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0812010147
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Autologous Stem Cell Transplant; ASCT; MM
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Dose Level 1 (Experimental): Dose Level 1; Bendamustine 30 mg/m^2 total, Melphalan 200 mg/m^2 total (140 mg/m^2 total for patients with Creatinine Clearance <70 ml/min)
  Interventions: Drug: Bendamustine; Drug: Melphalan
- Dose Level 2 (Experimental): Dose Level 2; Bendamustine 60 mg/m^2 total, Melphalan 200 mg/m^2 total (140 mg/m^2 total for patients with Creatinine Clearance <70 ml/min)
  Interventions: Drug: Melphalan; Drug: Bendamustine
- Dose Level 3 (Experimental): Dose Level 3; Bendamustine 90 mg/m^2 total, Melphalan 200 mg/m^2 total (140 mg/m^2 total for patients with Creatinine Clearance <70 ml/min)
  Interventions: Drug: Melphalan; Drug: Bendamustine
- Dose Level 4 (Experimental): Dose Level 4; Bendamustine 120 mg/m^2 total, Melphalan 200 mg/m^2 total (140 mg/m^2 total for patients with Creatinine Clearance <70 ml/min)
  Interventions: Drug: Melphalan; Drug: Bendamustine
- Dose Level 5 (Experimental): Dose Level 5; Bendamustine 150 mg/m^2 total, Melphalan 200 mg/m^2 total (140 mg/m^2 total for patients with Creatinine Clearance <70 ml/min)
  Interventions: Drug: Melphalan; Drug: Bendamustine
- Dose Level 6 (Experimental): Dose Level 6; Bendamustine 225 mg/m^2 total, Melphalan 200 mg/m^2 total (140 mg/m^2 total for patients with Creatinine Clearance <70 ml/min)
  Interventions: Drug: Melphalan; Drug: Bendamustine
- Phase 2 (Experimental): Bendamustine 225 mg/m^2 total, Melphalan 200 mg/m^2 total (140 mg/m^2 total for patients with Creatinine Clearance <70 ml/min)
  Interventions: Drug: Melphalan; Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — 30 mg/m^2 given on day 2 of melphalan
  Other Names: Treanda
  Arms: Dose Level 1
Drug: Melphalan — 100 mg/m^2 for 2 days (70 mg/m^2 for patients with Creatinine Clearance <70 ml/min)
  Other Names: Alkeran
Drug: Bendamustine — 60 mg/m^2 given on the 2nd day of melphalan
  Other Names: Treanda
  Arms: Dose Level 2
Drug: Bendamustine — 90 mg/m^2 given on the 2nd day of melphalan
  Other Names: Treanda
  Arms: Dose Level 3
Drug: Bendamustine — 60 mg/m^2 given on the 1st and 2nd day of melphalan
  Other Names: Treanda
  Arms: Dose Level 4
Drug: Bendamustine — 90 mg/m^2 given on the 1st day of melphalan and 60 mg/m^2 given on the 2nd day of melphalan
  Other Names: Treanda
  Arms: Dose Level 5
Drug: Bendamustine — 125 mg/m^2 given on the 1st day of melphalan and 100mg/m^2 given on the 2nd day of melphalan
  Other Names: Treanda
  Arms: Dose Level 6; Phase 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Bendamustine (TREANDA™), in combination with Melphalan in subjects with multiple myeloma who are undergoing an Autologous Stem Cell Transplant.

DETAILED DESCRIPTION:
Bendamustine (TREANDA™) has been used in clinical trials to treat multiple myeloma. The results from these trials suggest that it may be beneficial in the treatment of multiple myeloma in a different treatment context. Researchers aim to determine if there may be an improved benefit in the context of bone marrow transplant. This initial clinical trial is intended to help determine how safe it is to use bendamustine as a conditioning regimen for bone marrow transplant, and to look for any initial evidence of benefit.

Bendamustine (TREANDA™) is approved by the Food and Drug Administration (FDA) for the treatment of Chronic Lymphocytic Leukemia and Melphalan is a type of chemotherapy drug.

The use of Melphalan alone as a conditioning regimen for Autologous Stem Cell Transplant is considered "Standard of Care," that is, the treatment or process that your doctor would normally follow to treat your disease. Although Bendamustine (TREANDA™) has been used in multiple myeloma research studies, the combination of Bendamustine (TREANDA™) and Melphalan as treatment for Multiple Myeloma is not approved by the FDA, thus the combination therapy used in this research study is considered "investigational."

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma who have received induction therapy and have had stem cells mobilized in preparation for autologous transplantation will be eligible for this study. Patients are also eligible with relapsed or refractory disease, after attempts at more standard approaches, and with the availability of stem cells.
* Patients must be age 18 or older.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Patients must provide written informed consent.

Exclusion Criteria:

* Impaired renal function with a measured or calculated creatinine clearance of less than 25 ml/min.
* Impaired hepatic function defined as a bilirubin greater than 1.5 x upper limit of normal (ULN) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 5 x ULN.
* Serious active or uncontrolled infection or medical condition.
* Women who are pregnant or breast feeding. Women of childbearing age must use adequate contraception and have a negative pregnancy test.
* Impaired pulmonary function with a diffusing capacity of the lung for carbon monoxide (DLCO) less than 45% predicted.
* Impaired cardiac function with an ejection fraction less than 40% of predicted.
* Other systemic anticancer therapy or ongoing toxicities from such therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-04-23 (Actual); Primary Completion 2016-03-11 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsiporah Shore, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Derived] Gomez-Arteaga A, Mark TM, Guarneri D, Christos PJ, Gergis U, Greenberg JD, Hsu J, Mayer SA, Niesvizky R, Pearse RN, Phillips AA, Rossi A, Coleman M, van Besien K, Shore TB. High-dose bendamustine and melphalan conditioning for autologous stem cell transplantation for patients with multiple myeloma. Bone Marrow Transplant. 2019 Dec;54(12):2027-2038. doi: 10.1038/s41409-019-0587-0. Epub 2019 Jun 12. PMID 31190006

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four subjects were ineligible and therefore never started treatment.
Groups:
- Dose Level 1: Dose Level 1; Bendamustine 30 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
  Bendamustine: 30 mg/m2 given on day 2 of melphalan
  Melphalan: 100 mg/m2 for 2 days (70 mg/m2 for patients with Creatinine Clearance <70 ml/min)
- Dose Level 2: Dose Level 2; Bendamustine 60 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
  Melphalan: 100 mg/m2 for 2 days (70 mg/m2 for patients with Creatinine Clearance <70 ml/min)
  Bendamustine: 60 mg/m2 given on the 2nd day of melphalan
- Dose Level 3: Dose Level 3; Bendamustine 90 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
  Melphalan: 100 mg/m2 for 2 days (70 mg/m2 for patients with Creatinine Clearance <70 ml/min)
  Bendamustine: 90 mg/m2 given on the 2nd day of melphalan
- Dose Level 4: Dose Level 4; Bendamustine 120 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
  Melphalan: 100 mg/m2 for 2 days (70 mg/m2 for patients with Creatinine Clearance <70 ml/min)
  Bendamustine: 60 mg/m2 given on the 1st and 2nd day of melphalan
- Dose Level 5: Dose Level 5; Bendamustine 150 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
  Melphalan: 100 mg/m2 for 2 days (70 mg/m2 for patients with Creatinine Clearance <70 ml/min)
  Bendamustine: 90 mg/m2 given on the 1st day of melphalan and 60 mg/m2 given on the 2nd day of melphalan
- Dose Level 6: Dose Level 6; Bendamustine 225 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
  Melphalan: 100 mg/m2 for 2 days (70 mg/m2 for patients with Creatinine Clearance <70 ml/min)
  Bendamustine: 125 mg/m2 given on the 1st day of melphalan and 100mg/m2 given on the 2nd day of melphalan
- Phase 2: Bendamustine 225 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
  Melphalan: 100 mg/m2 for 2 days (70 mg/m2 for patients with Creatinine Clearance <70 ml/min)
  Bendamustine: 125 mg/m2 given on the 1st day of melphalan and 100mg/m2 given on the 2nd day of melphalan
Period: Phase 1
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Phase 2
Started | 3 | 6 | 3 | 3 | 3 | 8 | 0
Completed | 3 | 6 | 3 | 3 | 3 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Phase 2
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Phase 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 31
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 28
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1: Bendamustine 30 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
- Dose Level 2: Bendamustine 60 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
- Dose Level 3: Bendamustine 90 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
- Dose Level 4: Bendamustine 120 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
- Dose Level 5: Bendamustine 150 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
- Dose Level 6; Phase 2: Bendamustine 225 mg/m2 total, Melphalan 200 mg/m2 total (140 mg/m2 total for patients with Creatinine Clearance <70 ml/min)
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Phase 2 | Total
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 7 | 28 | 53
Age, Continuous [Median (Full Range); unit: years] | 56 [37 to 65] | 54.5 [46 to 62] | 58 [58 to 61] | 62 [62 to 65] | 53 [51 to 60] | 55 [48 to 66] | 61 [41 to 71] | 59 [37 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 1 | 4 | 15 | 26
  Male | 1 | 4 | 2 | 2 | 2 | 3 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 7
  Not Hispanic or Latino | 1 | 2 | 2 | 3 | 2 | 6 | 24 | 40
  Unknown or Not Reported | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 2 | 4 | 8
  White | 2 | 4 | 2 | 3 | 3 | 5 | 24 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (Phase 1)
Description: The Maximum Tolerated Dose was not met in Phase 1 of the study. Phase 2 participants were enrolled at the highest dose administered in Phase 1 (Dose Level 6) and this Outcome Measure is the reported number of dose-limiting toxicities experienced by Phase 1 participants. DLTs were defined as any grade 3 non-hematologic adverse even that did not resolve within 72 hours, any occurrence of a grade 4 non-hematologic adverse event, or failure to engraft with an absolute neutrophil count of 500/mm^3 and platelet count of 20,000/mm^3 untransfused by Day 35 post-transplant.
Time Frame: 35 days post-transplant
Population: Phase 1 includes all patients enrolled and treated on Phase 1 of the study (Dose Levels 1 through 6).
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: Dose Level 1; Bendamustine 30 mg/m^2 total, Melphalan 200 mg/m^2 total (140 mg/m^2 total for patients with Creatinine Clearance <70 ml/min)
  Bendamustine: 30 mg/m^2 given on day 2 of melphalan
  Melphalan: 100 mg/m^2 for 2 days (70 mg/m2 for patients with Creatinine Clearance <70 ml/min)
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 7
Participants | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Overall Response Rate (Phase 2) - Number of Participants Achieving at Least a Partial Response or Better in Disease Status at Day 100 Post-transplant
Description: Number of patients achieving at least a partial response or better in disease status at Day 100 post-transplant, as defined by the International Myeloma Working Group (IMWG) disease response criteria. Partial response in disease status is defined by the IMWG as ≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200 mg per 24 hours; If the serum and urine M-protein are unmeasurable, a ≥50% decrease in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria; If serum and urine M-protein are unmeasurable, and serum-free light assay is also unmeasurable, ≥50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma-cell percentage was ≥30%. In addition to these criteria, if present at baseline, a ≥50% reduction in the size (SPD) of soft tissue plasmacytomas is also required
Time Frame: 100 days post-transplant
Population: Phase 2 includes all patients treated on phase 2 of the study (28 patients), and patients treated at Dose Level 6 of the Phase 1 portion of the study (7 patients). The dose level used during Phase 2 was Dose Level 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 35
Participants | 33

3. Secondary Outcome: Progression-Free Survival (Phase 1)
Description: Time elapsed between Day 0 and disease progression, as defined by the International Myeloma Working Group (IMWG) disease response criteria. Disease progression is defined as an increase of >25% from lowest response value in any one or more of the following:
  * Serum M-component and/or (the absolute increase must be > 0.5 g/dL)
  * Urine M-component and/or (the absolute increase must be > 200 mg/24 h)
  * Only in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved free light chain levels. The absolute increase must be > 10 mg/dL
  * Bone marrow plasma cell percentage; the absolute percentage must be > 10%
  * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
  * Development of hypercalcaemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder
Time Frame: From Day 0 to first incidence of disease progression, up to 1,128 days
Population: Phase 1 includes all patients treated on Phase 1 of the study (Dose Levels 1-6). All cohorts were evaluated as one group for assessment of progression-free survival (PFS), as PFS is a secondary endpoint and there was no intent to stratify by cohort for the analysis. The number of patients per cohort is also too small for to evaluate by cohort.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Phase 1: Patients treated on Dose Level 1 through Dose Level 6. All patients received Melphalan 200 mg/m^2 total (140 mg/m^2 total for patients with Creatinine Clearance <70 ml/min).
  Dose Level 1; Bendamustine 30 mg/m^2 total Dose Level 2; Bendamustine 60 mg/m^2 total Dose Level 3; Bendamustine 90 mg/m^2 total Dose Level 4; Bendamustine 120 mg/m^2 total Dose Level 5; Bendamustine 150 mg/m^2 total Dose Level 6; Bendamustine 225 mg/m^2 total
Arm/Group | Phase 1
Number analyzed (Participants) | 25
Days | 791 [351 to NA] — Upper limit not estimable

4. Secondary Outcome: Progression-Free Survival (Phase 2)
Description: as for outcome 3
Time Frame: From Day 0 to first incidence of disease progression, up to 86 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2
Number analyzed (Participants) | 35
Months | 47 [34 to NA] — Upper limit was not estimable

5. Secondary Outcome: Overall Survival at 2 Years (Phase 1)
Description: Time elapsed between Day 0 and death from any cause, whichever came first, assessed up to 2 years.
Time Frame: From Day 0 until time of death, assessed up to 2 years.
Population: Phase 1 includes all patients treated on Phase 1 of the study (Dose Levels 1-6). All cohorts were evaluated as one group for assessment of overall survival, as overall survival is a secondary endpoint and there was no intent to stratify by cohort for the analysis. The number of patients per cohort is also too small for to evaluate by cohort.
Measure: Median (95% Confidence Interval); unit: Percentage of participants alive
Arm/Group | Phase 1
Number analyzed (Participants) | 25
Percentage of participants alive | 70 [43.9 to 85.7]

6. Secondary Outcome: Overall Survival at 3 Years (Phase 2)
Description: Time elapsed between Day 0 and death from any cause, whichever came first, assessed up to 3 years.
Time Frame: From Day 0 until time of death, assessed up to 3 years.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Percentage of participants alive
Arm/Group | Phase 2
Number analyzed (Participants) | 35
Percentage of participants alive | 88 [72 to 95]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed Day -2 through Day 100 post-transplant. All-Cause Morality was assessed for up to 2 years for Phase 2, and 3 years for Phase 2.
Description: All adverse events were first documented by the study transplant physicians and thereafter collated and graded by two independent reviewed according to CTCAE version 4.0.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Phase 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/6 | 0/3 | 0/3 | 1/3 | 1/7 | 6/28
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 0/3 | 0/3 | 0/3 | 0/7 | 8/28
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 3/3 | 3/3 | 7/7 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=6) | Dose Level 3 (N=3) | Dose Level 4 (N=3) | Dose Level 5 (N=3) | Dose Level 6 (N=7) | Phase 2 (N=28)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and Infestations - Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=6) | Dose Level 3 (N=3) | Dose Level 4 (N=3) | Dose Level 5 (N=3) | Dose Level 6 (N=7) | Phase 2 (N=28)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (13)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral Edema (Cardiac disorders) | 1 | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 13 (13)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (8)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (15)
Anorexia (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 2 (2) | 5 (5) | 12 (12)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 3 (3) | 3 (3) | 3 (3) | 5 (5) | 26 (26)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 20 (20)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Mucositis Oral (Gastrointestinal disorders) | 3 (3) | 6 (6) | 2 (2) | 3 (3) | 3 (3) | 6 (6) | 15 (15)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 7 (7) | 27 (27)
Rectal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 17 (17)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Fatigue (General disorders) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 27 (27)
Fever (General disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 7 (7)
Catheter-Related Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oral Thrush (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Alkaline Phopshatase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Weight Loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 26 (26)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 26 (26)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 10 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 10 (10)
Hypophospohatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 7 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 9 (9)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 8 (8)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 9 (9)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (5)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral Neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 10 (10)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 18 (18)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 14 (14)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 8 (8)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Rotavirus Enteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and Infestations - Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and Infestations - Streptococcus mitis Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and Infestations - Tinea pedia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and Infestations - Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and Infestations - Escherichia coli Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and Infestations - Clostridium difficile Colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and Infestations - Microsporidia Enteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Disorders - Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Nipple Sensitivity (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes